CLINICAL TRIAL: NCT07234552
Title: Impact of Abutment Screw Torque Values on Marginal Bone Loss and Peri-Implant Parameters: A Three-Arm Randomized Clinical Trial
Brief Title: Impact of Abutment Screw Torque on Marginal Bone Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan Carlos Bernabeu Mira, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-3792382
Record Dates: First submitted 2025-06-06; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Soft Tissues According to the Abutment Torque; Microleakage Accordint to the Abutment Torque; PROMS According to the Abutment Torque; Marginal Bone Loss According to the Abutment Torque
Keywords: Dental implant; Torque; Marginal bone loss; Microleakage; Abutment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transmucosal Abutment - 15 Ncm (Experimental)
  Interventions: Procedure: Abutment torqued to 15 Ncm
- Transmucosal Abutment - 30 Ncm (Experimental)
  Interventions: Procedure: Pilar torqued to 30 Ncm
- Submerged Healing Cap (No Transmucosal Connection) (Experimental)
  Interventions: Procedure: 2 mm healing cap

INTERVENTIONS:
Procedure: Abutment torqued to 15 Ncm — A dental implant surgery will be performed in which three implants will be placed. On one of them, a 2 mm slim abutment will be connected with a torque of 15 Ncm; on another, the same abutment will be connected with a torque of 30 Ncm; and on the third, a 2 mm healing cap will be placed and the implant will be left submerged for a subsequent second-stage surgery.
  Arms: Transmucosal Abutment - 15 Ncm
Procedure: Pilar torqued to 30 Ncm — A dental implant surgery will be performed in which three implants will be placed. On one of them, a 2 mm slim abutment will be connected with a torque of 15 Ncm; on another, the same abutment will be connected with a torque of 30 Ncm; and on the third, a 2 mm healing cap will be placed and the implant will be left submerged for a subsequent second-stage surgery.
  Arms: Transmucosal Abutment - 30 Ncm
Procedure: 2 mm healing cap — A dental implant surgery will be performed in which three implants will be placed. On one of them, a 2 mm slim abutment will be connected with a torque of 15 Ncm; on another, the same abutment will be connected with a torque of 30 Ncm; and on the third, a 2 mm healing cap will be placed and the implant will be left submerged for a subsequent second-stage surgery.
  Arms: Submerged Healing Cap (No Transmucosal Connection)

SUMMARY:
The objective of this clinical trial is to evaluate the impact of different torque values applied during transmucosal abutment placement in dental implants on marginal bone loss and peri-implant parameters, including the patient's perception of the treatment.

The main questions the study aims to answer are:

1. Is there any difference in marginal bone loss between abutments torqued at 15 Ncm, 30 Ncm, and submerged implants without immediate transmucosal connection?
2. Are there differences in microleakage between the different torque levels?
3. How do these torque values affect peri-implant soft tissues and patient satisfaction?
4. Does the applied torque influence the patient's quality of life after the prosthetic phase?

Each participant will receive three dental implants during the same surgical procedure. One of the following approaches will be applied to each implant:

1. A transmucosal abutment torqued to 15 Ncm
2. A transmucosal abutment torqued to 30 Ncm
3. A healing cap without transmucosal connection (submerged implant)

After implant placement, clinical and radiographic assessments will be performed to measure marginal bone loss and peri-implant parameters.

DETAILED DESCRIPTION:
This study aims to analyze how different torque levels applied during transmucosal abutment placement on dental implants influence peri-implant tissue health and other relevant clinical parameters. A randomized clinical trial will be conducted in which each participant will receive three dental implants. Each implant will be assigned to one of the following conditions: an abutment torqued to 15 Ncm, an abutment torqued to 30 Ncm, and a submerged implant with a healing cap, without immediate transmucosal connection.

This intra-individual design enables direct comparison of outcomes while minimizing inter-individual variability that could affect the results.

Throughout the treatment process, various data will be collected. During surgery, patient-reported comfort levels will be recorded. Following prosthesis placement, standard clinical measurements will be performed, including peri-implant probing, bleeding on probing, inflammation, and radiographic evaluation of marginal bone loss.

Additionally, patient-reported outcomes during the first week after the initiation of the prosthetic phase will be documented, including pain levels, inflammation, and analgesic use. Overall satisfaction and the impact of treatment on quality of life will also be assessed using a Likert-type scale, focusing on functions such as chewing, speech, sleep, and daily activities.

The goal of this study is to determine whether the torque applied during abutment connection has a clinically relevant effect on both peri-implant tissue response and patient perception of the treatment. The findings may contribute to improved clinical guidelines in implant dentistry and enhance long-term treatment outcomes.

The study protocol has been approved by the relevant ethics committee and will comply with all applicable clinical research regulations. All participants will provide written informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Posterior edentulism
* Completion of craniofacial growth
* Full-mouth plaque index and bleeding index < 25%
* Sufficient bone height and width for implant placement without the need for bone regeneration procedures
* Presence of at least 2 mm of keratinized mucosa around the dental implant
* Stable occlusion and healthy periodontium
* Absence of medical conditions that contraindicate implant surgery, such as heavy smoking (<10 cigarettes per day), severe bruxism, pregnancy or breastfeeding, bisphosphonate therapy, and patients undergoing chemotherapy or radiotherapy in the head and/or neck area
* Uncooperative patients

Exclusion Criteria:

* Loss to follow-up
* Incorrectly parallelized periapical radiographs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss (mm) assessed by standardized periapical radiographs | Day 0 (surgery); 1 month post-op; 3 months post-op (prosthetic loading); and 1, 3, 6, and 12 months post-loading. Unit of measure: Milimeters (mm)
  Marginal bone loss will be measured on standardized digital periapical radiographs taken using the parallel technique. A calibrated digital tool will be used to determine the vertical distance from the implant-abutment junction to the most coronal bone-to-implant contact on the mesial and distal sides. Measurements will be collected at seven time points for each participant.

SECONDARY OUTCOMES:
Postoperative pain intensity (VAS) | Immediately after surgery; 1, 3, and 7 days post-surgery; and 1, 3, and 7 days post-loading. Unit of measure: Points on a 0-10 scale
  Pain intensity will be evaluated using a 10-point Visual Analog Scale (VAS), where 0 represents "no pain" and 10 represents "worst imaginable pain." Participants will complete the VAS at specified time points following surgery and prosthetic loading. Higher scores indicate more intense pain.
  This measure is part of the Patient-Reported Outcome Measures (PROMs) evaluated in this study.
Postoperative swelling (VAS) | Immediately after surgery; 1, 3, and 7 days post-surgery; and 1, 3, and 7 days post-loading. Unit of measure: Points on a 0-10 scale
  Facial swelling will be assessed using a 10-point Visual Analog Scale (VAS), where 0 represents "no swelling" and 10 represents "severe swelling." Assessments will be recorded at defined postoperative intervals. Higher scores indicate greater swelling.
  This measure is part of the Patient-Reported Outcome Measures (PROMs) evaluated in this study.
Patient satisfaction with surgical and prosthetic phases (Likert-type questionnaire) | 1 month post-op (surgical phase) and 3 months post-op (prosthetic loading). Unit of measure: Points on a likert-type scale
  Satisfaction with the surgical and prosthetic phases will be assessed using Likert-type questionnaires addressing comfort, duration, and overall perception. Higher scores indicate greater satisfaction.
  This measure is part of the Patient-Reported Outcome Measures (PROMs) evaluated in this study.
Oral health-related quality of life (Likert-type questionnaire) | Baseline (before surgery); 1 month post-op; and 12 months post-loading. Unit of measure: Points on a likerts-type scale
  Oral health-related quality of life-including speech, chewing, sleep, mouth opening, work, daily routine, and analgesic intake-will be assessed using Likert-type questionnaires. Higher scores indicate greater quality-of-life impact.
  This measure is part of the Patient-Reported Outcome Measures (PROMs) evaluated in this study.
Peri-implant probing depth (mm) | 3 months post-op (prosthetic loading); and 1, 3, 6, and 12 months post-loading. Unit of measure: Milimeters (mm)
  Probing depth will be measured at four sites per implant (mesial, distal, buccal, lingual) using a calibrated periodontal probe. The mean value per implant will be recorded. Lower values indicate healthier peri-implant tissues.
Bleeding on probing (presence/absence) | 3 months post-op (prosthetic loading); and 1, 3, 6, and 12 months post-loading. Unit of measure: Percentage of implant sites with bleeding (%)
  Bleeding on probing will be assessed at four sites per implant (mesial, distal, buccal, lingual). The presence or absence of bleeding within 30 seconds after gentle probing will be recorded. The percentage of sites showing bleeding will be calculated for each implant. Lower percentages indicate healthier peri-implant tissues.
Mucosal inflammation (visual assessment) | 3 months post-op (prosthetic loading); and 1, 3, 6, and 12 months post-loading. Unit of measure: Presence or absence of inflammation (binary)
  Mucosal inflammation around each implant will be evaluated by visual inspection for redness, swelling, and other clinical signs. Each implant site will be classified as showing inflammation or not. Lower prevalence of inflammation indicates healthier peri-implant tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Claver Baldovi, Principal Investigator — University of Valencia

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) has not yet been determined. A final decision will depend on data quality, ethical considerations, and publication status.